CLINICAL TRIAL: NCT04978142
Title: Transcranial Modulation of Oscillatory Brain Activity in People With Tinnitus: A Concurrent Transcranial Direct Current Stimulation (tDCS) - Magnetoencephalography (MEG) Study
Brief Title: MaST: MEG and Brain Stimulation in Tinnitus
Acronym: MaST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Magdalena Sereda, Senior Research Fellow, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 505-2003
Record Dates: First submitted 2021-06-29; First posted 2021-07-27 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Active tDCS stimulation at 2 mA for 20 minutes, with a 10 seconds of ramp-up and 10 seconds of ramp-down time as used in previous tinnitus studies. The stimulation will be delivered via two rubber electrodes attached using a layer of conductive paste (35 cm2). The anode will be placed over the right dlPFC and cathode over the left dlPFC).
  Interventions: Device: transcranial Direct Current Stimulation (tDCS)
- Sham (Sham Comparator): Placebo stimulation is performed using the same current intensity, but only applied for 45 seconds in addition to the 10 second ramp-up and 10 second ramp-down periods. The electrode configuration and placement will be identical to the active stimulation.
  Interventions: Device: transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: transcranial Direct Current Stimulation (tDCS) — Non-invasive neuromodulation employing a direct current, applied using a DC STIMULATOR PLUS manufactured by NeuroConn Technology by NeuroCare. This is a micro-processor-controlled constant current source. It meets the highest safety standards thanks to (hardware- and software-based) multistage monitoring of the current path. By continuously monitoring electrode impedance it can detect insufficient contact with the skin and automatically terminate stimulation. This is a reliable method of avoiding any injury to the patient.

SUMMARY:
Tinnitus is the awareness of a sound in the ear or head without any outside source. It affects around 15% of people in the UK. About 20% of people with tinnitus experience symptoms that negatively affect their quality of life including sleep disturbances, difficulties with hearing and concentration, social isolation, anxiety, depression, irritation or stress. Most common clinical management strategies for tinnitus include education and advice combined with some form of sound therapy. The effects of these management options are, however, variable. Currently, the exact aetiology of tinnitus is unknown although maladaptive plasticity due to sensorineural hearing loss is thought to play a big role. Neuroimaging studies have pointed to over-activation or excessive spontaneous activity within the central auditory cortex. Furthermore, electrophysiological techniques have confirmed the frontal cortex's role in tinnitus through dysfunctional top-down modulation.

Transcranial direct current stimulation (tDCS) is a neurostimulation technique in which weak currents (1-2 mA's) are delivered to the brain, thereby depolarising or hyperpolarising neurons within the desired region of cortex. tDCS is a non-invasive and easy to apply tool, delivered by applying two surface electrode to a patients head. It has previously been used as a treatment for depression, stroke rehabilitation, and cognitive enhancement.

Some studies have indicated potential benefit of tDCS in tinnitus patients, but this has not yet been investigated within the UK. Neuromodulation therapies should deliver a permanent reduction in tinnitus percept by driving the neuroplastic changes necessary to interrupt abnormal levels of oscillatory cortical activity and restore typical levels of activity. This change in activity should alter or interrupt the tinnitus percept (reduce or extinguish) and this should be concomitant with a change in the level of self-reported tinnitus handicap. The currently ongoing Cochrane review of neuromodulation (desynchronisation) for tinnitus in adults found mixed evidence for the electrical stimulation therapies for tinnitus, including tDCS. However, the review also found that the most recent tDCS trials that have used greater numbers of treatment sessions found significant reductions in tinnitus symptom severity, anxiety, and depression. Authors concluded that these findings warrant further trials of tDCS. Research studies using electroencephalography (EEG) or magnetoencephalography (MEG) suggested changes in oscillatory activity in different frequency bands that might be associated with tinnitus, however a consistent picture has not yet emerged. Reduction of this abnormal activity might signify a reduction in the level or perceived severity of TI and could potentially be used as a valuable indicator of the course of TI treatment.

In this project specific changes in brain activity that happen during a new treatment approach for tinnitus - transcranial Direct Current Stimulation (tDCS)- will be investigated. This will help to determine how the treatment might work, whether specific brain activity may be a meaningful biological indicator or objective measure of tinnitus, and provide a reliable measure of treatment-related change; this has not yet been achieved in tinnitus research but is crucial.

DETAILED DESCRIPTION:
Data collection session will involve the participant completing the Tinnitus Functional Index (TFI) and Demographics and Tinnitus History Questionnaire (D&THQ), which will provide the investigators with information about their personal tinnitus history including subjective characteristics such as loudness. The D&THQ consists of questions selected from the European School for Interdisciplinary Tinnitus Research Screening Questionnaire (ESIT-SQ). Participants will undergo a standard hearing test, which will inform the investigators of any hearing loss. The participant's head shape will be digitized to aid in the spatial localization of the MEG signal. The participant will then undergo 40 minutes of MEG scanning (10 minutes of resting state without tDCS, 20 minutes of resting state MEG with either active or sham tDCS, and then another 10 minutes of resting state MEG without tDCS. The first 10 minutes will serve as a baseline of resting state oscillatory brain activity. The concurrent tDCS and MEG recording will allow the investigators to observe changes in oscillatory brain activity during tDCS. The last 10 minutes of MEG recording will allow the investigators to see whether any changes in oscillatory activity persist after the stimulation ends. After the MEG recording has finished, the participant will undergo an anatomical MRI scan. This will allow the investigators to take the participants' individual brain morphology into account when analysing the source of the MEG signal.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or over
2. Have subjective tinnitus
3. Able to read and understand English
4. Safe to undergo tDCS (according to tDCS Safety Questionnaire)
5. Safe to undergo MRI scanning (according to MRI Safety Screening Questionnaire)

Exclusion Criteria:

1. Aged under 18 years
2. No tinnitus
3. Not able to read and understand English
4. Not safe to undergo tDCS (according to tDCS Safety Questionnaire)
5. Not safe to undergo MRI scanning (according to MRI Safety Screening Questionnaire)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Oscillatory activity | Continuously for 10 minutes before the onset of the intervention, continuously for 20 minutes before the intervention, continuously for 10 minutes after the intervention
  Change in oscillatory resting state activity as measured with magnetoencephalography (MEG)
Connectivity | Continuously for 10 minutes before the onset of the intervention, continuously for 20 minutes before the intervention, continuously for 10 minutes after the intervention
  Change in functional neural connectivity as measured with magnetoencephalography (MEG)
Tinnitus loudness | Within 5 minutes after intervention
  Loudness of tinnitus percept as measured by visual analogue scale (0-10) with a higher score meaning louder tinnitus

SECONDARY OUTCOMES:
Blinding | Within 5 minutes after intervention
  Effectiveness of blinding using a questionnaire
Adverse effects | Within 5 minutes after intervention
  Type and severity of adverse effects measured with adverse affects questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena N Sereda, PhD, Principal Investigator — NIHR Nottingham BRC / University of Nottingham; Bas Labree, MSc, Study Director — NIHR Nottingham BRC / University of Nottingham
Locations (1):
- University of Nottingham, NIHR Nottingham Biomedical Research Centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adjamian P, Sereda M, Hall DA. The mechanisms of tinnitus: perspectives from human functional neuroimaging. Hear Res. 2009 Jul;253(1-2):15-31. doi: 10.1016/j.heares.2009.04.001. Epub 2009 Apr 11. PMID 19364527
- [Background] Adjamian P, Sereda M, Zobay O, Hall DA, Palmer AR. Neuromagnetic indicators of tinnitus and tinnitus masking in patients with and without hearing loss. J Assoc Res Otolaryngol. 2012 Oct;13(5):715-31. doi: 10.1007/s10162-012-0340-5. Epub 2012 Jul 12. PMID 22791191
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Genitsaridi E, Partyka M, Gallus S, Lopez-Escamez JA, Schecklmann M, Mielczarek M, Trpchevska N, Santacruz JL, Schoisswohl S, Riha C, Lourenco M, Biswas R, Liyanage N, Cederroth CR, Perez-Carpena P, Devos J, Fuller T, Edvall NK, Hellberg MP, D'Antonio A, Gerevini S, Sereda M, Rein A, Kypraios T, Hoare DJ, Londero A, Pryss R, Schlee W, Hall DA. Standardised profiling for tinnitus research: The European School for Interdisciplinary Tinnitus Research Screening Questionnaire (ESIT-SQ). Hear Res. 2019 Jun;377:353-359. doi: 10.1016/j.heares.2019.02.017. Epub 2019 Mar 2. PMID 30871820
- [Background] Faber M, Vanneste S, Fregni F, De Ridder D. Top down prefrontal affective modulation of tinnitus with multiple sessions of tDCS of dorsolateral prefrontal cortex. Brain Stimul. 2012 Oct;5(4):492-8. doi: 10.1016/j.brs.2011.09.003. Epub 2011 Oct 5. PMID 22019079
- [Background] Yadollahpour A, Mayo M, Saki N, Rashidi S, Bayat A. A chronic protocol of bilateral transcranial direct current stimulation over auditory cortex for tinnitus treatment: Dataset from a double-blinded randomized controlled trial. F1000Res. 2018 Jun 12;7:733. doi: 10.12688/f1000research.14971.1. eCollection 2018. PMID 30356442